CLINICAL TRIAL: NCT03764722
Title: Effectiveness of a Repetitive Use of 24-hour Levosimendan Infusions in Patients With Severe Systolic Heart Failure in Order to Prevent Rehospitalizations
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Collegium Medicum w Bydgoszczy (Other)
Responsible Party: Principal Investigator, Małgorzata Dobosiewicz, PhD, Professor Grzegorz Grześk, Collegium Medicum w Bydgoszczy
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KB 431/2018
Record Dates: First submitted 2018-07-26; First posted 2018-12-05 (Actual); Last update posted 2018-12-05 (Actual); Status verified 2018-12

CONDITIONS: Systolic Heart Failure
Keywords: Levosimendan; Rehospitalisation; Heart failure
MeSH Terms: conditions — Heart Failure, Systolic; Heart Failure | interventions — Simendan

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Levosimendan (Experimental)
  Interventions: Drug: Levosimendan

INTERVENTIONS:
Drug: Levosimendan — The patient will initially receive a standard dose of 0.1 mcg/kgmc/min. In case of good tolerance of the drug - the dose will be increased to 0.2 mcg/kgmc/min. If hypotension SBP <90 mmHg occurs, the dose will be reduced to 0.05 mcg / kgm / min. If the hypotension persists despite the reduction of the drug - the infusion will be terminated and the patient will be excluded from the study. The infusion will be terminated within 24 hours, the patient will be examined again 4 hours after the end of the infusion, by the attending physician and unless there are contraindications - discharged home.
  Patients will be hospitalized every 4 weeks for the next 6 months.

SUMMARY:
Rehospitalizations due to exacerbation of chronic heart failure are an important problem for patients suffering from heart failure.

Rehospitalzations lead to worse prognosis, have an impact on the quality of life and have a negative financial impact on the health care system.

Currently, studies are being conducted on the efficacy of levosimendan in the prevention of heart failure exacerbations. Patients receive levosimendan at repetitive use and preliminary results suggest a reduction in the incidence of exacerbations of heart failure.

Thanks to the clinical trial planned in the Department of Cardiology of the Biziel Hospital with repeatable use of levosimendan, it is possible to determine the benefits of this method of treatment more accurately.

DETAILED DESCRIPTION:
Heart failure affects 12% of the adult population and its frequency increases with age and affects 10% of people over 70 years old. Heart failure is characterized by high annual death rate reaching 17% and the percentage of rehospitalization at the level of 44% annually. In order to reduce morbidity and mortality rates in the case of heart failure, many diagnostic and therapeutic methods have been introduced over the last few years, however the prognosis for this medical condition is still unfavorable nonetheless.

Rehospitalizations due to exacerbation of chronic heart failure are an important problem for patients suffering from heart failure.

Rehospitalzations lead to worse prognosis, have an impact on the quality of life and have a negative financial impact on the health care system. At the moment, there are numerous clinical trials aimed at improving the prognosis of patients with heart failure.

Levosimendan is a modern drug registered in the treatment of acute heart failure. In the current ESC guidelines for the treatment of patients with acute heart failure, levosimendan is mainly recommended for the group of patients chronically treated with beta-adrenolytics and in the treatment of a peri-infarction shock.

It is a substance with inotropic positive and vasodilating effects. It belongs to the group of drugs sensitizing contractile elements of a myocardium on calcium ions. In the clinical trials and meta-analyses, the safety profile of levosimendan is better in comparison to the classical pressure amines used in the treatment of acute heart failure: dobutamine and dopamine. Beneficial clinical effect of levosimendan is prolonged beyond the period of its direct use due to the active metabolites remaining in the bloodstream.

Currently, studies are being conducted on the efficacy of levosimendan in the prevention of heart failure exacerbations. Patients receive levosimendan at repetitive use and preliminary results suggest a reduction in the incidence of exacerbations of heart failure. Due to the low number of patients included in individual centers and non-homogeneous protocols of the use of levosimendan in repeated infusions, the benefits of using this method of treatment can not be clearly determined at present. Thanks to the clinical trial planned in the Department of Cardiology of the Biziel Hospital with repeatable use of levosimendan, it is possible to determine the benefits of this method of treatment more accurately.

Levosimendan is a drug with a beneficial safety profile, and the most common side effect, which is hypotension, will disappear shortly after discontinuation of treatment or after an infusion of crystalloids. Patients will be hospitalized at ITK, where a standard physical examination will be conducted. The patient will fill in the SF36 questionnaire before the treatment to self-evaluate his or hers quality of life. The patient will take medication according to the latest outpatient recommendations.

During the 24-hour treatment, blood pressure will be monitored (until the target dose is set). The heart rate will be monitored continuously (for the next 2 hours every 30 minutes, then every 1 hour). Daily balance of fluids will be administered.

The patient will initially receive a standard dose of 0.1 mcg/kgmc/min. In case of good tolerance of the drug - the dose will be increased to 0.2 mcg/kgmc/min. If hypotension SBP <90 mmHg occurs, the dose will be reduced to 0.05 mcg / kgm / min. If the hypotension persists despite the reduction of the drug - the infusion will be terminated and the patient will be excluded from the study. The infusion will be terminated within 24 hours, the patient will be examined again 4 hours after the end of the infusion, by the attending physician and unless there are contraindications - discharged home.

Patients will be hospitalized every 4 weeks for the next 6 months with the above-mentioned parameters from the peripheral blood and march test, before the next dose. The control test will also include the determination of the concentration of levosimendan metabolites prior to the next infusion.

During the last follow-up visit, echocardiography and spiroergometry testing will be performed before the next dosage.

After the 12 months of inclusion in the study, a telephone interview will be conducted in the direction of rehospitalization due to exacerbation of heart failure.

The data obtained from the study will be compared with the standard parameters of rehospitalization due to the exacerbation of heart failure included in the ESC guidelines. The variability of data obtained from the quality of life questionnaire at the beginning and at the end of the study will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

- at least 2 hospitalizations due to exacerbation of chronic heart failure with reduction of left ventricular ejection fraction (EF< 40%) during last 6 months, despite optimal heart failure treatment

Exclusion Criteria:

* chronic kidney disease (GFR < 30)
* severe liver damage (AT 5x > N, bilirubin >2,0 g/dl)
* hypotonia
* hypokalemia
* HGB<10g/dl
* severe aortic and mitral stenosis
* tachycardia >100/min or atrial fibrillation with HR > 120/min
* features of hypovolemia
* levosimendan intolerance
* acute infection

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of rehospitalisations in patients with severe heart failure treated with 24-hour levosimendan infusions | 12 months

SECONDARY OUTCOMES:
Change in quality of life in patients with severe heart failure treated with 24-hour levosimendan infusions. | from baseline up to 4 weeks during 6 months
  via SF-36 questionnaire
Change in sodium in patients with severe heart failure treated with 24-hour: SF-36 questionnaire levosimendan infusions. | from baseline up to 4 weeks during 6 months
  counted in mmol/l
Change in kaldyum in patients with severe heart failure treated with 24-hour levosimendan infusions. | from baseline up to 4 weeks during 6 months
  counted in mmol/l
Change in NT-proBNP in patients with severe heart failure treated with 24-hour levosimendan infusions. | from baseline and up to 4 weeks during 6 months.
  counted in ng/l
Change in troponin T in patients with severe heart failure treated with 24-hour levosimendan infusions. | from baseline and up to 4 weeks during 6 months.
  counted in μg/l

CONTACTS AND LOCATIONS:
Overall Officials: Grzegorz Grześk, Professor, Principal Investigator — Collegium Medicum w Bydgoszczy
Locations (1):
- Second Department of Cardiology, Bydgoszcz, Poland

IPD SHARING:
Plan to Share IPD: No